CLINICAL TRIAL: NCT06715761
Title: Effectiveness of Manual and Instrumental Myofascial Release in Chronic Low Back Pain and the Posture of Practitioners CrossFit®: Protocol of a Randomized Controlled Clinical
Brief Title: Effectiveness of Manual and Instrumental Myofascial Release in Chronic Low Back Pain and the Posture of Practitioners CrossFit®
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gabriela Souza de Vasconcelos (Other)
Responsible Party: Sponsor-Investigator, Gabriela Souza de Vasconcelos, Professor, Universidade Federal de Goias
Organization: Universidade Federal de Goias (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Federal University of Goiás
Record Dates: First submitted 2024-11-13; First posted 2024-12-04 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Low Back Pain
Keywords: Low back pain; Myofascial release; CrossFit; Posture
MeSH Terms: conditions — Low Back Pain | interventions — Myofascial Release Therapy; Cupping Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Myofascial release group (MRG) (Experimental)
  Interventions: Other: Myofascial release
- Cupping therapy group (CTG) (Active Comparator)
  Interventions: Other: Cupping therapy
- Control group (CG) (No Intervention): Wait-and-see

INTERVENTIONS:
Other: Myofascial release — The sequence of myofascial release is as follows: 30 seconds of contact between the therapist's hands and the entire region of the participant's spine, sliding with medium pressure in a caudocranial direction; palpation of the erector spinae, quadratus lumborum, gluteus and piriformis muscles bilaterally, to identify trigger points, marking each point of tension with a dermographic pencil for subsequent manipulation; 3 cycles of bilateral paravertebral release, by sustained pressure with crossed hands, until the restrictive tissue barrier is found, for 60 seconds; 90 seconds of the vertical rolling technique (superficial elevation of the skin and mobilisation of the tissue with the tips of all the fingers) on the bilateral paravertebrals and, at the end, sliding along the entire length of the bilateral multifidus, with the fingers flexed, using the bony prominence between the proximal and middle phalanges as contact with the skin, in a caudocranial direction and returning craniocaudal.
  Arms: Myofascial release group (MRG)
Other: Cupping therapy — The acrylic cups (DongBang®) will be placed on the meridional points, as Traditional Chinese Medicine calls them, 1 cup in the central region of each popliteal fossa, the so-called B40 or Wei Zhong point, 6 cups in the region of the quadratus lumborum muscles, more specifically on the BL23 or Shenshu points (approximately 5 centimetres lateral to the edge of the L2 spinous process), BL24 or Qihaishu (approximately 5 centimetres lateral to the edge of the spinous process of L3) and BL25 or Dachangshu (approximately 5 centimetres lateral to the edge of the spinous process of L4) bilaterally, as well as a cup on a single point of the participant's choice, where they report the most lower back pain (ashi point). The cups will be attached to the skin using a gun, applying two suction pressures, and the participant will be asked to signal whether the pressure is strong or weak. The cups will remain attached for 12 minutes on the B40 meridian and 15 minutes on the other meridians. If a cup lo
  Arms: Cupping therapy group (CTG)

SUMMARY:
Background: Chronic low back pain (LBP) can lead to major functional disabilities and force people to take time off work, sports or leisure activities. Regular physical exercise is an important ally in reducing the risk factors for most diseases, and CrossFit® is one of the modalities that has been gaining momentum when choosing an exercise. However, the intensity recommended in training can collaborate with the development of musculoskeletal problems such as pain and postural changes, interfering with the development of the practice, with low back pain being one of the most common disorders in these practitioners, especially caused by mechanical stress. Considering that CrossFit® practitioners have already incorporated physical exercise into their routine, passive techniques such as myofascial release (ML) have been discussed as a form of treatment for LBP. For this reason, this study was designed to verify the efficacy of ML in the LBP of CrossFit® practitioners, comprising two techniques, one manual and one instrumental, and to see if the outcome of the LBP alters the posture of the spine.

This is a randomised controlled clinical that will be conducted in a CrossFit® box in the city of Goiânia-GO, Brazil. At least 51 people will take part who have been doing CrossFit® for at least 3 months, who have LBP, are aged between 18-59 and are not undergoing any other treatment for low back pain. There will be two experimental groups, one that will receive manual MR and the other, cupping therapy, as well as a control group that will not receive any technique. The sessions will take place twice a week for 8 weeks. The primary outcome will be low back pain intensity, assessed at baseline, weekly and after 8 weeks, and the secondary outcomes, which will be postural deviations, spinal mobility and history of musculoskeletal pain, assessed at baseline and at the end of 8 weeks. There will be no blinding between therapist and participants.

Discussion: This study will investigate whether MR is effective in relation to LBP, given that some results have already shown positive responses in acute conditions, while also verifying the repercussions on the postural aspect. The results could provide additional knowledge about the best technique to use and, having applicability to our outcomes, will favour and simplify treatment, helping professionals to make clinical decisions.

ELIGIBILITY:
Inclusion Criteria:

* men and women aged between 18 and 59 years;
* presence of low back pain for at least 12 weeks;
* have started regular CrossFit® activity at least 3 months ago.

Exclusion Criteria:

* perform other physical activity than CrossFit®;
* continuous use of painkillers;
* previous pathologies or spinal surgery;
* amputations;
* haematological disorders;
* fibromyalgia;
* hypersensitivity or skin lesions.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Baseline, once a week throughout the intervention period (at the beginning of each week) and post intervention (8 weeks)
  Pain intensity, related to chronic low back pain, will be measured using the Visual Analogue Scale (VAS), where 0 represents "no pain" and 10 represents "the worst pain possible". Participants will indicate their usual pain.

SECONDARY OUTCOMES:
Spinal postural deviations | Baseline and post intervention (8 weeks)
  Spinal postural deviations will be measured using a flexible lead ruler called a Flexicurve (Trident®). Initially, the anatomical points of the spinous processes of the C7, T1, T6, T12, L1, L4, L5, S1 and S2 vertebrae will be marked on the participant's skin with a white dermatographic pencil (Hintz®). The flexicurve will then be moulded and the anatomical reference points will also be marked on the body of the ruler. After this, the ruler will be positioned in the centre of the page of a 420mmX549mm piece of graph paper (Tracing Pad®), where its shape will be reproduced. For the analysis, the drawings with the shapes of the curvatures of the spine will be photographed and entered into the Dynamic Posture software.
Spine mobility | Baseline and post intervention (8 weeks)
  Spinal mobility will be analysed using Finger Tip Test. For the Finger Tip Test, the participant will stand and then be instructed to flex their trunk as if they wanted to touch their hands to the floor. The distance between the distal phalanx of the 3rd finger of the hand and the floor will be measured with a tape measure (Incoterm®).
History of musculoskeletal pain | Baseline and post intervention (8 weeks)
  A history of musculoskeletal pain will be taken using the Questionnaire For Evaluation Of Musculoskeletal Pain In Exercise Practitioners (Q-ADOM). The questionnaire is used to screen for musculoskeletal pain in exercise practitioners and, although it has domains that can cover any type of pain, the participant will be instructed to answer the visual analogue scale (item 1) and the other items, only considering the intensity of the pain and the symptoms related to their chronic low back pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Goias, Goiânia, Goiás, Brazil

IPD SHARING:
Plan to Share IPD: No